CLINICAL TRIAL: NCT03386799
Title: Evaluation of a Power Assistance Device for Wheelchair-DUO
Acronym: EVALDUO
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_75; 2017-A02670-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Paraplegia; Hemiplegia
Keywords: Power assistance device; Wheelchair
MeSH Terms: conditions — Paraplegia; Hemiplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient in wheelchair: Patient in wheelchair with E-motion device
  Interventions: Device: E-motion device

INTERVENTIONS:
Device: E-motion device — Powered assisted Wheelchair with the E-motion device. Outdoor and indoor runs

SUMMARY:
Power assisted wheelchairs have specific advantages compared to manual propelled or powered Wheelchair. Autonomad Mobility has developed a new device (DUO), the assistance being triggered by the motion of the wheelchair and not an push on the hand rim, people who use their foot to move or people pushing the wheelchair can be helped by the device as people propelling the wheelchair with their arms.

Furthermore DUO has an option with a longer assistance (AEP+) which can be preferred by some people.

To be referenced and reimbursed by the French health insurance, DUO has to be compared with an other power assistance device for wheelchairs, already referenced.

The study is a comparative study between DUO and the ALBER E Motion. Each patient is his own control and is assessed in 4 experimental conditions, with intervals of 3 or 4 days, manually propelled, with the E mtion device, with the DUO device and the single push configuration, with the DUO device and the AEP+ configuration.

The main outcome measure will be the user's satisfaction (using 8 items of the ESAT questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* with a motor deficiency (of any origin) needing a manual wheelchair
* propelling his wheelchair with both arms or with one foot and one arm.
* covered by the French national health insurance.
* living at less than 30km form the investigation center

Exclusion Criteria:

* subject of a guardianship or tutelage measure
* owning already a power wheelchair or a powered assisted wheelchair
* with cognitive impairments that affect the steering capacity or the understanding of the instructions.
* Patient unable to use a manual wheelchair indoor without help,
* Contraindication in keeping a seating position especially the occurrence of ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a motor deficiency (of any origin) needing a manual wheelchair
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
ESAT questionnaire | at 12 days
  User satisfaction, using 8 items of the ESAT (Echelle de Satisfaction envers une Aide Technique) questionnaire

SECONDARY OUTCOMES:
Success rate during the indoor test (wheelchair skill program) | at 12 days
Time to perform the wheelchair skill program | at 12 days
Time run | at 12 days
  During a 500 m outdoor run
Maximal heart rate | at 12 days
  During a 500 m outdoor run
Effort assessment by the Borg scale | at 12 days
  During a 500 m outdoor run The 10-point Borg scale ranges from 0 "nothing at all" to 10 "maximal/extremely strong" and will be used to rate the intensity of dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: André Thevenon, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedauw, CHU, Lille, France